CLINICAL TRIAL: NCT06611254
Title: Quantification of Brain and Kidney Perfusion Before, During, and After Hypothermia Treatment in Neonates With Perinatal Asphyxia Using Contrast-enhanced Ultrasound
Status: Recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Ferdinand Knieling, Principal Investigator, Pediatric Translational Imaging Laboratory, University of Erlangen-Nürnberg Medical School
Other Study IDs: Neo_CEUS_ULM
Record Dates: First submitted 2024-06-21; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Perinatal Asphyxia; Hypothermia Treatment; Gestational Age Min. 36SSW

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates with perinatal asphyxia and indication for hypothermia treatment: Included will be neonates with perinatal asphyxia that get an indication for hypothermia treatment (severe azidosis and signs of encephalopathy and under 6h of age and >36 gest. weeks). They will be monitored with CEUS/ULM at three different time points (T1: within first 6h of life/before hypothermia treatment, T2 = during hypothermia treatment/6-78h of life, T3 = after hypothermia treatment/within first week of life.
  Interventions: Device: Contrast enhanced ultrasound imaging (CEUS) and post processing with ULM

INTERVENTIONS:
Device: Contrast enhanced ultrasound imaging (CEUS) and post processing with ULM — CEUS is a contrast based ultrasound technique and ULM (Ultrasound Localization Microscopy) is a post-processing bioinformatical method to quantify microvascular architecture and perfusion dynamics.

SUMMARY:
In this clinical study vascular dynamics in the neonatal brain and kidney will be monitored by CUES and ULM before, during and after hypothermia treatment in neonates with asphyxia.

DETAILED DESCRIPTION:
Perinatal asphyxia (PA) is the reduced supply of oxygen to vital organs during or immediately after birth. PA is one of the most common causes of neonatal mortality in full-term infants worldwide and of hypoxic-ischemic encephalopathy (HIE) with subsequent neurological deficits (spastic cerebral palsy). In addition to brain damage, perinatal asphyxia often leads to dysfunction of other organs. It is not uncommon for this to be accompanied by transient renal failure.

Hypothermia treatment is an established therapeutic measure for neuroprotection in clinical indications of HIE. This involves lowering the core body temperature of affected children to 33.5°C for 72 hours. The therapeutic effect is thought to be due to multifactorial mechanisms, including a reduction in endothelial dysfunction, reduced excretion of free radicals and attenuation of the inflammatory cascade.

In the guidelines for hypothermia treatment in neonatal asphyxia, regular ultrasound examinations are prescribed to clarify damage to the central nervous system (CNS) before, during and after hypothermia treatment.1 In infants, transfontal ultrasound makes it possible to visualize brain structures, vessels and their flow velocities.

The intravenous use of ultrasound contrast enhancers as an aid also opens up the possibility of recording the tissue perfusion of the CNS and kidneys, including the smallest vessels.8 This could provide significantly more information compared to conventional methods and expand our knowledge of the pathophysiology and individual status of tissue perfusion in patients.

For example, two studies at Erlangen University Hospital have successfully used contrast-enhanced ultrasound (CEUS) with the contrast agent known as SonoVue® to visualize postoperative perfusion of the brain after pediatric cardiac surgery.

In this clinical study, the new CEUS measurement and imaging technique will be used before, during and after hypothermia treatment in neonates with asphyxia. A contrast agent (SonoVue®) will be administered during the routine ultrasound examination and improved tissue visualization will be achieved. The aim is to gain new insights into brain and kidney perfusion as part of the treatment and to better assess the extent of organ damage in the individual patient through more specific vascular imaging. Improved visualization and assessment of the end-stream area will provide information on processes that promote the development of HIE and renal failure. Finally, the aim is to compare diagnostic and prognostic methods with the currently recommended measures. The CEUS is to be examined as a possible diagnostic imaging tool and possibly a supplement to existing diagnostic methods.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of the inclusion criteria for hypothermia treatment according to the AWMF guideline
* Severe acidosis (pH ≤7.0 or a base deficit ≥16 mmol/l) in umbilical cord blood or a blood sample from the first hour of life, and
* clinical signs of moderate or severe encephalopathy (severity grade 2 or 3 according to Sarnat & Sarnat), and
* postnatal age ≤6h, and
* gestational age ≥36 weeks' gestation
* Consent of the parents/legal guardians
* Time 1 (before the start of hypothermia treatment)

  * Informing the parents/legal guardians present on site despite an emotionally stressful situation with high individual benefit for the patient
  * If only one parent is present and able to provide information, their consent is sufficient - the second parent is informed repeatedly when they regain the ability to provide information
  * Information adapted to the emergency situation, addressing the personal situation and comprehensible presentation of the plan
* Time 2 (during hypothermia treatment)

  -->Offer of a further informative discussion/repeated explanation with the parents/legal representatives before the second measurement in order to answer any questions that may have arisen
* Suitable acoustic window
* Availability of the qualified examiner

Exclusion Criteria:

* Lack of consent of at least one parent
* Pre-existing brain malformations
* Absence of the competent examiner

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: One study population. Anticipated approx. n=20 neonateswith above mentioned inclusion criteria with perinatal asphyxia and inclusion criteria for hypothermia treatmentaccording to the AWMF guideline.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
CEUS Time intensity curves | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  All CEUS outcomes will be generated in order to achieve time intensity curves in contrast enhanced ultrasound analysis
CEUS Measurement1 | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  PE (Peak-Enhancement)
CEUS Measurement2 | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  WiAUC (Wash-in Area Under the Curve (AUC(TI: TTP)))
CEUS Measurement3 | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  WiAUC (Wash-in Area Under the Curve (AUC(TI: TTP)))
CEUS Measurement4 | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  RT (Rise Time)
CEUS Measurement5 | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  mTT (mean Transit Time local) (mTT-TI))
CEUS Measurement6 | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  TTP (Time to Peak)
CEUS Measurement7 | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  WiR (Wash-in-Rate )
CEUS Measurement8 | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  WiPI (Wash-in Perfusion Index (WiAUC/RT))
CEUS Measurement9 | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  WoAUC (Wash-out AUC (AUC(TTP:TO)))
CEUS Measurement10 | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  WiWoAUC (Wash-in- und Wash-out-AUC (WiAUC+WoAUC))
CEUS Measurement11 | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  FT (Fall Time - (TO-TTP))
CEUS Measurement12 | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  WOR (Wash-out-Rate) QOF (Quality Of Fit between the echo-power signal and f(t)
CEUS Measurement13 | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  QOF (Quality Of Fit between the echo-power signal and f(t)
Near-infrared spectroscopy | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  Near-infrared spectroscopy Non-invasive measurement of oxygen saturation in tissue using a probe that is attached to the head.62 This procedure is already firmly established in the field of pediatric surgery and pediatric cardiology interventions at the University Hospital Erlangen. The probe is attached before the start of the first measurement time point and removed after the end of the third measurement time point. There is no risk of side effects.
Visualization and quantification of cerebral perfusion with CEUS | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  CEUS imaging for cerebral perfusion in asphyxia
Visualization and quantification of of renal perfusion with CEUS | before(T1, within the first 6hours of life), during hypothermia treatment(T2, 6-78hours of life), after treatment (T3, within first week of life)
  CEUS imaging for renal perfusion in asphyxia

SECONDARY OUTCOMES:
CEUS and NIRS | T1,T2,T3
  Correlation coefficient (R) between CEUS curve and NIRS
Neurological status assessment (Bayley Score) | Month of life: 3-4 and 6-24
  Neurological status of the patients will be assessed by the score "Bayley Scales of Infant and Toddler Development"
MRI imaging in asphyxia | once within first two years of life
  MRI Weeke Score
Comparison of the CEUS time-intensity curve between three timepoints | T1,T2, T3
  CEUS curve at T1,T2, T3
Assessment of blood Lactate | T1, T2, T3
  Lactate (mmol/l)
EEG signs of seizures | T1 -T3 and through study completion
  Number (n) of ETPs in EEG
EEG activity | T1 -T3 and through study completion
  frequency EEG (Hz)
Assessment of renal function GFR | T1 -T3 and through study completion, an average of 3 years
  GFR (ml/min/1,73 m2)
Assessment of renal function urea | T1 -T3 and through study completion, an average of 3 years
  urea (mg/dl)
Assessment of renal function urinary status | T1 -T3 and through study completion
  standardized urinary status
Assesment of renal function kreatininekinase | T1, T2, T3
  kreatininekinase (U/l)
Assessment of metabolic LDH | T1, T2, T3
  LDH (U/l)

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Knieling, MD, Principal Investigator — FAU Erlangen-Nuernberg; Gregor Hanslik, MD, Principal Investigator — FAU Erlangen-Nuernberg
Locations (1):
- FAU Erlangen-Nuernberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No